CLINICAL TRIAL: NCT00760929
Title: A Randomized, Placebo Controlled Study to Determine the Effect of Two Dose Schedules of R1507 or Placebo, Both in Combination With Erlotinib (Tarceva®), on Progression-free Survival in Patients With Advanced Non-small Cell Lung Cancer With Disease Progression After First or Second Line Chemotherapy
Brief Title: A Study of the Effect of R1507 in Combination With Tarceva (Erlotinib) on Progression-Free Survival in Patients With Stage IIIb/IV Non-Small Cell Lung Cancer (NSCLC).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to the termination of the clinical development program.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NO21160; 2008-001736-12 (EudraCT Number)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — RG-1507 monoclonal antibody; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo for R1507 (16mg/kg iv) (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: erlotinib [Tarceva]
- Placebo for R1507 (9mg/kg iv) (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: erlotinib [Tarceva]
- R1507 (16mg/kg iv) (Experimental)
  Interventions: Drug: RG1507; Drug: erlotinib [Tarceva]
- R1507 (9mg/kg iv) (Experimental)
  Interventions: Drug: RG1507; Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: Placebo — iv 9mg/kg weekly
  Arms: Placebo for R1507 (9mg/kg iv)
Drug: Placebo — iv 16mg/kg every 3 weeks
  Arms: Placebo for R1507 (16mg/kg iv)
Drug: RG1507 — iv 9mg/kg weekly
  Arms: R1507 (9mg/kg iv)
Drug: RG1507 — iv 16mg/kg every 3 weeks
  Arms: R1507 (16mg/kg iv)
Drug: erlotinib [Tarceva] — 150mg oral daily

SUMMARY:
This 4 arm study in patients with advanced Stage IIIb/IV non-small cell cancer (NSCLC) who failed at least one standard chemotherapy regimen will determine the proportion of patients with progression-free survival at 12 weeks following combination therapy with R1507 and Tarceva or placebo and Tarceva. Patients will be randomized to one of four treatment arms to receive R1507 (9mg/kg iv) or placebo weekly or R1507 (16mg/kg iv) or placebo every 3 weeks. Tarceva (150mg oral daily) will be administered in all treatment arms. Other disease-related endpoints including overall survival, objective response rate, time to response, time to progressive disease and duration of response will also be evaluated. The anticipated time on study treatment is 1-2 years, and the target sample size is <500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients >=18 years with histologically documented inoperable, locally advanced or metastatic (stage IIIB or IV) NSCLC;
* patients must have failed at least one but no more than two standard chemotherapy regimens;
* measurable disease according to the RECIST criteria;
* Eastern Cooperative Oncology Group (ECOG) performance status;
* life expectancy >12 weeks.

Exclusion Criteria:

* patients with active central nervous system (CNS) lesions;
* prior treatment with agents acting via insulin-like growth factor 1 receptor (IGF-1R) inhibition or epidermal growth factor receptor (EGFR) targeting;
* administration with high doses of systemic corticosteroids;
* radiotherapy in the 4 weeks prior to study start;
* surgery or significant traumatic injury with in the last 2 weeks prior to study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2008-11-10 (Actual); Primary Completion 2010-06-25 (Actual); Study Completion 2010-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (57):
- United States (15):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Florida Cancer Inst., New Port Richey, Florida
  - Emory Univ Winship Cancer Inst, Atlanta, Georgia
  - University of Chicago Medical Center; Dept. of Medicine/Section of Nephrology, Chicago, Illinois
  - North Shore University Health System, Glenview, Illinois
  - Joliet Oncology Hematology Associates, Ltd., Joliet, Illinois
  - St. Joseph Medical Center, Towson, Maryland
  - Massachusetts General Hospital., Boston, Massachusetts
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Carolina Oncology Specialists, PA - Hickory, Hickory, North Carolina
  - Chattanooga Oncology and Hematology Associates, PC, Chattanooga, Tennessee
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - Virginia Cancer Institute, Richmond, Virginia
- Australia (3):
  - Flinders Medical Center; Medical Oncology, Adelaide, South Australia
  - Frankston Hospital; Oncology/Haematology, Frankston, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (5):
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Notre Dame, Charleroi
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven
  - Chr de La Citadelle, Liège
- Lakeridge Health Oshawa; Oncology, Oshawa, Ontario, Canada
- France (5):
  - Hopital Albert Michallon; Medecine Aigue Specialisee Pneumologie, La Tronche
  - Hopital de La Croix Rousse; Service de Pneumologie, Lyon
  - Fondation Hopital Saint Joseph; Pole Cancerologie, Imagerie Medicale Service d'Oncologie, Paris
  - Hopital Tenon;Pneumologie, Paris
  - Hopital Larrey; Clinique Des Voies Respiratoires, Toulouse
- Germany (9):
  - Zentralklinik Bad Berka GmbH; Pneumologie, Bad Berka
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH; Klinik fuer Innere Medizin I, Halle
  - Asklepios Klinik Harburg; Thoraxzentrum, Hamburg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Stiftung Kathol. Krankenhaus Marienhospital Herne Klinik Mitte Frauenklinik, Herne
  - Klinikum Leverkusen; Med. Klinik III / Onkologie, Leverkusen
  - Ludwig-Maximilians Uni Klinik Innenstadt; Medizinische Klinik, München
- St. James Hospital; Oncology, Dublin, Ireland
- Italy (5):
  - Arcispedale Santa Maria Nuova; Oncologia, Reggio Emilia, Emilia-Romagna
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Az. Osp. S. Luigi Gonzaga; Malattie Apparato Respiratorio 5 Ad Indirizzo Oncologico, Orbassano, Piedmont
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; Oncologia Medica, Sant'Andrea Delle Fratte (PG), Umbria
- Poland (4):
  - Medical University of Gdansk, Gdansk
  - SK Przemienienia Panskiego UM im.K.Marcinkowskiego, Poznan
  - Specjalistyczny Szpital Im. Prof. A. Sokolowskiego; Oddziall Chemioterapii, Szczecin
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
- Spain (5):
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Majadahonda, Madrid
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga
- United Kingdom (4):
  - Royal Surrey County Hospital; St. Lukes Cancer Centre, Guildford
  - Wythenshawe Hospital; North West Lung Centre, Manchester
  - Sir Bobby Robson Cancer Research Centre, Newcastle upon Tyne
  - New Cross Hospital; Deansley Centre, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Ramalingam SS, Spigel DR, Chen D, Steins MB, Engelman JA, Schneider CP, Novello S, Eberhardt WE, Crino L, Habben K, Liu L, Janne PA, Brownstein CM, Reck M. Randomized phase II study of erlotinib in combination with placebo or R1507, a monoclonal antibody to insulin-like growth factor-1 receptor, for advanced-stage non-small-cell lung cancer. J Clin Oncol. 2011 Dec 1;29(34):4574-80. doi: 10.1200/JCO.2011.36.6799. Epub 2011 Oct 24. PMID 22025157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A screening examination was to be performed between -28 and 1 days before first day of treatment.
Pre-assignment Details: Safety population was used for the participant flow. All randomized participants who received at least one treatment. Two patients randomized to placebo QW actually received R1507 9 mg/kg QW.
Groups:
- Placebo for R1507 (9mg/kg iv): Participants received a placebo equivalent to R1507 (9mg/kg iv) intravenously every week until disease progression.
- Placebo for R1507 (16mg/kg iv): Participants received the placebo equivalent to R1507 (16 mg/kg iv) intravenously every 3 weeks until disease progression.
- R1507 (9mg/kg iv): Participants received R1507 (9mg/kg iv) intravenously every week until disease progression.
- R1507 (16mg/kg iv): Participants received R1507 (16 mg/kg iv) intravenously every 3 weeks until disease progression.
Period: Overall Study
Arm/Group | Placebo for R1507 (9mg/kg iv) | Placebo for R1507 (16mg/kg iv) | R1507 (9mg/kg iv) | R1507 (16mg/kg iv)
Started | 26 | 29 | 59 | 57
Completed | 0 | 1 | 1 | 2
Not Completed | 26 | 28 | 58 | 55
Not completed — Adverse Event | 2 | 0 | 6 | 10
Not completed — Lack of Efficacy | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 9 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Progression of Disease | 21 | 26 | 38 | 42
Not completed — Other | 2 | 0 | 2 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Violation of Selection Criteria at Entry | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population was used for the baseline population. All randomized participants who received at least one treatment. Two patients randomized to placebo QW actually received R1507 9 mg/kg QW.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo for R1507 (9mg/kg iv) | Placebo for R1507 (16mg/kg iv) | R1507 (9mg/kg iv) | R1507 (16mg/kg iv) | Total
Number analyzed (Participants) | 26 | 29 | 59 | 57 | 171
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (8.01) | 62.3 (8.26) | 60.3 (10.45) | 60.5 (9.82) | 61.0 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 18 | 19 | 57
  Male | 17 | 18 | 41 | 38 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 0 | 1 | 1 | 1 | 3
  Hispanic | 0 | 1 | 1 | 0 | 2
  White | 26 | 27 | 57 | 56 | 166
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 3 | 6 | 8 | 5 | 22
  Never smoked | 3 | 4 | 6 | 7 | 20
  Past smoker | 20 | 19 | 45 | 45 | 129

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS)
Description: PFS was defined as the time at which half of the participants have progressed (progressive disease [PD]) based on RECIST tumor response criteria or died from any cause, whichever occurred first. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Participants who had not died or progressed at the time of the final analysis were censored at the date of last contact.
Time Frame: 12 weeks
Population: All-treated population: All participants enrolled in the study who had been randomly assigned to one of the four study treatments were included. For analysis, participants receiving both weekly and every 3 weeks of placebo were combined and evaluated as one group.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received a placebo equivalent to R1507 (9mg/kg iv) intravenously every week until disease progression or the placebo equivalent to R1507 (16 mg/kg iv) intravenously every 3 weeks until disease progression.
Arm/Group | Placebo | R1507 (9mg/kg iv) | R1507 (16mg/kg iv)
Number analyzed (Participants) | 57 | 57 | 57
Participants
  Progression-Free & Alive | 18 | 16 | 21
  Progressed, Died, or Unknown | 39 | 41 | 36

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the median time, in weeks, from the date of randomization to the date of death, due to any cause. Participants who have not died at the time of the final analysis will be censored at the date the participant was last known to be alive. The 90% CI was estimated using Kaplan-Meier methodology.
Time Frame: From baseline up to 20 months
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Placebo | R1507 (9mg/kg iv) | R1507 (16mg/kg iv)
Number analyzed (Participants) | 57 | 57 | 57
Weeks | 35.1 [20.9 to 44.7] | 35.1 [26.1 to 43.4] | 52.4 [33.7 to 65.7]
Statistical Analysis 1: Comparison: Placebo vs R1507 (9mg/kg iv); Test type: Superiority; p = 0.4301, Wald Test; Hazard Ratio (HR) = 0.84, 90% CI [0.58 to 1.21]
Statistical Analysis 2: Comparison: Placebo vs R1507 (16mg/kg iv); Test type: Superiority; p = 0.0342, Wald Test; Hazard Ratio (HR) = 0.61, 90% CI [0.42 to 0.90]

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) was defined by RECIST criteria as the best response achieved by a patient over the course of the trial, which includes a complete response (CR) or partial response (PR) that has been confirmed by a second tumor assessment no earlier than 4 weeks after the initial documentation, stable disease (SD), or progressive disease (PD). PR was defined as ≥ 30% decrease in sum of longest diameter of all target lesions, from baseline sum. CR was defined as disappearance of all target and non-target lesions. For CR or PR, tumor measurements must be confirmed by 2nd assessments within 4 weeks. PD = 20% increase in the sum of longest diameter of all target lesions, from smallest sum of longest diameter of all target lesions recorded at or after baseline; or a new lesion; or progression of non-target lesions. SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on the study.
Time Frame: From baseline up to 20 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | R1507 (9mg/kg iv) | R1507 (16mg/kg iv)
Number analyzed (Participants) | 57 | 57 | 57
Percentage of Participants | 8.8 [3.5 to 17.6] | 7 [2.4 to 15.3] | 7 [2.4 to 15.3]

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the first documented complete response (CR) or partial response (PR) to the first documented disease progression (PD) or death, whichever occurs first. A CR was defined as the disappearance of all target lesions (TL). A PR was defined as at least a 30% decrease in the sum of the longest diameter (SLD) of TLs taking as reference the Baseline SLD. PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since treatment started or the unequivocal progression of existing non-TLs.
Time Frame: From baseline up to 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | R1507 (9mg/kg iv) | R1507 (16mg/kg iv)
Number analyzed (Participants) | 5 | 4 | 4
days | 260.40 (140.56) | 215.50 (91.70) | 257.75 (130.07)

5. Secondary Outcome: Time to Response
Description: This is defined for participants with objective response, as the date of randomization to the date of first CR or PR which will be the date the response is first radiographically documented following initiation of therapy (the date of the actual imaging modality).
Time Frame: From baseline up to 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | R1507 (9mg/kg iv) | R1507 (16mg/kg iv)
Number analyzed (Participants) | 5 | 4 | 4
days | 42.40 (4.34) | 65.25 (22.95) | 85.25 (34.70)

ADVERSE EVENTS:
Time Frame: Baseline up to 20 months
Description: Multiple occurrences of the same adverse event in one individual counted only once. Safety population was used for the participant flow. All randomized participants who received at least one treatment. Two patients randomized to placebo QW actually received R1507 9 mg/kg QW.
Arm/Group | Placebo for R1507 (9mg/kg iv) | Placebo for R1507 (16mg/kg iv) | R1507 (9mg/kg iv) | R1507 (16mg/kg iv)
All-Cause Mortality (participants affected / at risk) | 20/26 | 22/29 | 43/59 | 34/57
Serious Adverse Events (participants affected / at risk) | 5/26 | 3/29 | 18/59 | 14/57
Other Adverse Events (participants affected / at risk) | 26/26 | 27/29 | 57/59 | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo for R1507 (9mg/kg iv) (N=26) | Placebo for R1507 (16mg/kg iv) (N=29) | R1507 (9mg/kg iv) (N=59) | R1507 (16mg/kg iv) (N=57)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 (0) | 1 (1) | 1 (1)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 (0) | 1 (1) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERITONITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo for R1507 (9mg/kg iv) (N=26) | Placebo for R1507 (16mg/kg iv) (N=29) | R1507 (9mg/kg iv) (N=59) | R1507 (16mg/kg iv) (N=57)
RASH (Skin and subcutaneous tissue disorders) | 14 (14) | 16 (16) | 32 (32) | 42 (42)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 5 (5) | 7 (7)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 5 (5) | 4 (4)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
ACNE (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 10 (10) | 13 (13) | 30 (30) | 32 (32)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 4 (4) | 20 (20) | 19 (19)
VOMITING (Gastrointestinal disorders) | 6 (6) | 5 (5) | 14 (14) | 7 (7)
STOMATITIS (Gastrointestinal disorders) | 3 (3) | 3 (3) | 9 (9) | 15 (15)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 1 (1) | 9 (9) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (6) | 7 (7)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
FATIGUE (General disorders) | 4 (4) | 7 (7) | 22 (22) | 23 (23)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 4 (4) | 7 (7) | 11 (11)
ASTHENIA (General disorders) | 6 (6) | 2 (2) | 10 (10) | 2 (2)
PYREXIA (General disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 8 (8) | 10 (10)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 9 (9) | 10 (10)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 10 (10) | 12 (12)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (4)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
PARONYCHIA (Infections and infestations) | 0 (0) | 2 (2) | 5 (5) | 5 (5)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 6 (6) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 2 (2)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 2 (2) | 2 (2) | 7 (7) | 6 (6)
DIZZINESS (Nervous system disorders) | 4 (4) | 3 (3) | 5 (5) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 6 (6)
PARAESTHESIA (Nervous system disorders) | 3 (12) | 1 (3) | 2 (3) | 1 (2)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (4) | 8 (8) | 13 (13) | 22 (22)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (4) | 1 (1) | 3 (3) | 5 (5)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 8 (8) | 12 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 1 (1) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 6 (6) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 1 (1) | 15 (15) | 9 (9)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
DEPRESSION (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 4 (4) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Development of the study drug R1570 was discontinued based on the available clinical data and the large number of molecules targeting the pathway. Not all efficacy parameters described in the protocol were assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.